CLINICAL TRIAL: NCT04198259
Title: Interventional Devascularization Plus HVPG-Guided Carvedilol Therapy vs TIPS for the Prevention of Gastric Variceal Rebleeding in Patients With Liver Cirrhosis: A Prospective, Randomized, Controlled Trial
Brief Title: Interventional Devascularization Plus HVPG-Guided Carvedilol Therapy vs TIPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Tie Jun, Director of clinical research, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY20192116-F-1
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Gastric Varices Bleeding; Liver Cirrhoses
Keywords: TIPS; HVPG; BRTO; NSBB
MeSH Terms: interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional devascularization (Active Comparator): Interventional devascularization includes BRTO and similar procedure. Several variations of the technique exist, such as balloon-occluded antegrade transvenous obliteration or occlusion of the collateral by the placement of a vascular plug or coils.
  Interventions: Procedure: interventional devascularization
- Transjugular intrahepatic portosystemic shunt (Experimental): TIPS is an artificial channel within the liver that establishes communication between the inflow portal vein and the outflow hepatic vein.
  Interventions: Procedure: TIPS

INTERVENTIONS:
Procedure: interventional devascularization — Interventional devascularization (BRTO and its variations) is a procedure for treatment of fundal varices associated with a large gastro-/splenorenal collateral.
  Arms: interventional devascularization
Procedure: TIPS — TIPS is very effective in the treatment of bleeding GV, with more than a 90% success rate for initial hemostasis. It frequently requires additional embolization of spontaneous collaterals feeding the varices. The incidence of encephalopathy was higher after TIPS.
  Arms: Transjugular intrahepatic portosystemic shunt

SUMMARY:
Gastric varices (GV) are present in around 20% of patients with cirrhosis. Bleeding from GV accounts for 10-20% of all variceal bleeding. For the prevention of gastric variceal bleeding, TIPS or BRTO as firstline treatments were suggested.

No randomized trials have compared BRTO with other therapies. BRTO and its variations might increase portal pressure and might worsen complications, such as ascites or bleeding from EV. In this regard, if NSBB is combined with BRTO and its variations (we called interventional devascularization) for those HVPG responders, the drawbacks of interventional devascularization might be overcome. Therefore, the investigators conducted this RCT to compare the effectiveness and safety of TIPS with those of interventional devascularization in the prevention of rebleeding from gastric varices.

DETAILED DESCRIPTION:
Gastric varices (GV) are present in around 20% of patients with cirrhosis. Bleeding from GV accounts for 10-20% of all variceal bleeding. GV are classified according to their location in the stomach and their relationship with esophageal varices (EV). Accordingly, GV are divided into gastroesophageal varices (GOV) and isolated gastric varices (IGV) . The management of type 1 GOV, which extend from the esophagus along the lesser curvature of the stomach, is similar to the management of EV. Historically, bleeding from type 2 GOV (i.e. GOV extending into the fundus), type 1 IGV (i.e. located in the fundus) and type 2 IGV (i.e. located anywhere in the stomach), is considered to be more severe and difficult to treat than EV bleeding. Few studies, mostly retrospective and uncontrolled, have focused on the management of non-GOV1 GV, and the optimal treatment remains controversial.

For the prevention of gastric variceal bleeding, treatment principles can be classified into two categories: decreasing portal pressure and obstructing GEV. Methods for decreasing portal pressure include medications (NSBB), radiological intervention (TIPS) and surgery. In contrast, methods for treating the obstruction of GEV include endoscopic approaches (EVL, EIS) or radiological intervention (such as BRTO). Recent portal hypertensive bleeding suggested TIPS or BRTO as firstline treatments in the prevention of rebleeding.

BRTO is a procedure for treatment of fundal varices associated with a large gastro-/splenorenal collateral. The technique involves retrograde cannulation of the left renal vein by the jugular or femoral vein, followed by balloon occlusion and slow infusion of sclerosant to obliterate the gastro-/splenorenal collateral and fundal varices. Several variations of the technique exist, such as balloon-occluded antegrade transvenous obliteration or occlusion of the collateral by the placement of a vascular plug or coils. BRTO has the theoretical advantage over TIPS that it does not divert portal blood inflow from the liver. On the other hand, BRTO and its variations might increase portal pressure and might worsen complications, such as ascites or bleeding from EV. In this regard, if NSBB is combined with BRTO and its variations (we called interventional devascularization) for those HVPG responders, the drawbacks of interventional devascularization might be overcome.

Therefore, the investigators conducted this RCT to compare the effectiveness and safety of TIPS with those of interventional devascularization in the prevention of rebleeding from gastric varices.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis diagnosed by clinical examination, imaging or biopsy
* Patients with a previous history of variceal hemorrhage
* Gastric variceal confirmed by an endoscopic examination, including IGV1 or IGV2
* Aged 18 to 75 years
* Adequate liver and kidney function, including Child-Turcotte-Pugh score < 12, MELD score <19, and serum creatinine less than 2 times the upper limit of normal.

Exclusion Criteria:

* Active variceal bleeding
* Esophageal variceal, including GOV1 or GOV2 type, mainly esophageal varices;
* Refractory ascites
* Patients with contraindication to treatment of TIPS, including congestive heart failure, NYHA III and IV, pulmonary arterial hypertension(>50mmHg), polycystic liver, intrahepatic duct dilatation, spontaneous bacterial peritonitis, hepatic encephalopathy
* Patients with contraindication to treatment of Carvedilol, including asthma, insulin-dependent diabetes, peripheral vascular diseases
* Child-Turcotte-Pugh score >=12, or MELD score >=19
* Budd-Chiari syndrome
* The main portal vein thrombosis is greater than 50%
* Malignancies
* An uncontrolled infection
* Previously treated with TIPS, splenectomy pericardia vascular disconnection, or surgical shunts
* HIV or HIV related illness
* Allergic to contrast agent
* Lactating or pregnant
* Non-compliant patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of gastric variceal rebleeding | 12 months
  Confirmed by endoscopy

SECONDARY OUTCOMES:
Cumulative incidence of variceal hemorrhage related death | 12 months
Cumulative incidence of hepatic encephalopathy (HE) | 12 months
  HE is classified as covert HE and overt HE
Cumulative incidence of death | 12 months
  all cause mortality
Cumulative incidence of adverse events | 12 months
  number of adverse events and adverse reactions in each arm
Correlation between hepatic venous pressure gradient response and cardiac index response to Carvedilol | 12 months
  Investigate non-invasive tools for risk stratification

CONTACTS AND LOCATIONS:
Overall Officials: Jun Tie, M.D.,Ph.D., Principal Investigator — Air Force Military Medical University, China